CLINICAL TRIAL: NCT03791957
Title: The Association of the Levels of Blood Haemoglobin to the Distribution and Severity of Gingival Melanin Pigmentation at 3 Different Periodontal Health Status
Brief Title: The Association of Blood Haemoglobin and Colour of Gums
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr. Riya Achamma Daniel, Post graduate student, Principal investigator, Department of Periodontics, KLE Society's Institute of Dental Sciences, Bangalore, KLE Society's Institute of Dental Sciences
Other Study IDs: riya2pigmentation
Record Dates: First submitted 2018-12-30; First posted 2019-01-03 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Gingival Pigmentation; Gingivitis; Periodontitis; Healthy
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A - Healthy Periodontium: Absence of clinical signs of inflammation like bleeding on probing, erythema, edema, attachment loss, bone loss, patient symptoms, (bone levels at 1-3mm apical to CEJ) n=20
  Interventions: Other: Blood Haemoglobin
- Group B - Gingivitis: Presence of cardinal signs of inflammation along with, bleeding and discomfort on gentle probing, loss of knife-edged margin and blunting of papilla, n=20
  Interventions: Other: Blood Haemoglobin
- Group C - Periodontitis: Presence of cardinal signs of inflammation along with, bleeding and discomfort on gentle probing, loss of knife-edged margin and blunting of papilla,periodontal pocketing, clinical attachment loss, radiographically assessed bone loss n=20
  Interventions: Other: Blood Haemoglobin

INTERVENTIONS:
Other: Blood Haemoglobin — Routine haemotological investigation of blood haemoglobin levels in gm/dL will be recorded from withdrawn venous blood

SUMMARY:
AIM:

To evaluate the association of the levels of blood haemoglobin to the distribution and severity of gingival melanin pigmentation at 3 different periodontal health status

SAMPLE SIZE ESTIMATION

* Done using GPower v.3.1.9.2
* Total sample size = 60 (20 each in 3 groups)
* Effect size = 40%
* Power = 80%
* α-error = 5%

SAMPLING:

* Simple random sampling
* Subjects to be recruited from out patient pool of KLE Society's Institute of Dental Sciences, Bangalore
* Subjects to be categorised into 3 groups (20 subjects each)

  1. Group A - Healthy periodontium
  2. Group B - Gingivitis
  3. Group C - Periodontitis

PARAMETERS ASSESSED

* Blood Haemoglobin Concentration (in %gm/dL)
* Hedin Melanin Index Score 0: No pigmentation Score 1: one or two solitary unit(s) of pigmentation in papillary gingiva without formation of a continuous ribbon between solitary units Score 2: More than three units of pigmentation in papillary gingiva without the formation of a continuous ribbons of pigmentation Score 3: One or more short continuous ribbons of pigmentation Score 4: One continuous ribbon including the entire area between canines

STATISTICAL ANALYSIS

* SPSS for Windows Version 22.0 to be used
* Descriptive statistics: It includes expression of study parameters in terms of Mean & SD for continuous variables, whereas in terms of frequency and proportions for categorical variables.
* Inferential Statistics:

Chi Square Test will be used to compare the pigmentation index between 03 groups. And similarly, gender wise comparison of hemoglobin concentration will be done using the same test.

One-way ANOVA test followed by Tukey's HSD post hoc Analysis will be used to compare the mean hemoglobin levels based on the pigmentation index scores in each group.

The level of significance [P-Value] was set at P<0.05

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Absence of pathological gingival pigmentation

  1. Group A - Healthy Periodontium: Absence of clinical signs of inflammation like bleeding on probing, erythema, edema, attachment loss, bone loss, patient symptoms, (bone levels at 1-3mm apical to CEJ)
  2. Group B - Gingivitis: Presence of cardinal signs of inflammation along with, bleeding and discomfort on gentle probing, loss of knife-edged margin and blunting of papilla,
  3. Group C - Periodontitis: Presence of cardinal signs of inflammation along with, bleeding and discomfort on gentle probing, loss of knife-edged margin and blunting of papilla,periodontal pocketing, clinical attachment loss, radiographically assessed bone loss

Exclusion Criteria:

* Tobacco associated pigmentation - smoker's melanosis, chewing/ pouching tobacco
* Pigmentation from exogenous pigments - amalgam tattoo, cultural tattooing, beverages, food colours, betelnut/khat chewing, heavy metals ( mercury, silver, arsenic, bismuth, graphite, lead), topical medications, other foreign bodies
* Pigmentation from endogenous pigments - jaundice, ecchymosis/ petechiae, haemochromatosis, hemosiderin
* Long term consumption of pigmentation causing drugs - ACTH, antimalarial drugs, busulfan, doxorubicin, minocycline, oral contraceptives, phenothiazies
* Syndromes and systemic diseases associated with pigmentation - Addison's disease. Albright's syndrome, basila melanosis, β-thalassemia, healed / healing mucocutaneous lesions, hereditary hemorrhagic Telangiectasia, HIV-associated melanosis, Neurofibromatosis, Peutz Jeghers syndrome, hamartoma, pyogenic granuloma, epulis
* Benign or malignant lesions involving gingival - angiosarcoma, hemangioma, Kaposi's sarcoma, malignant melanoma, melanocytic nevus, pigmented vaculoe

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects to be recruited from out patient pool of KLE Society's Institute of Dental Sciences, Bangalore, India
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Blood Haemoglobin to Melanin pigmentation | Baseline
  To assess the association of the levels of blood haemoglobin to the distribution and severity of gingival melanin pigmentation at 3 different periodontal health status by Hedin Melanin Index both by intragroup comparison within each of the 3 groups and intergroup comparison between the three groups

IPD SHARING:
Plan to Share IPD: No